CLINICAL TRIAL: NCT02227589
Title: Treatment for Teens With Alcohol Abuse and Depression
Acronym: T-TAAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: UConn Health (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00053448; 1R01AA021719-01A1 (NIH); 1R01AA021735-01A1 (NIH)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2019-02

CONDITIONS: AOD Use, Abuse, and Dependence; Depression
Keywords: adolescent,; alcohol abuse; depression,; cognitive behavior therapy; cannabis abuse
MeSH Terms: conditions — Depression; Alcoholism; Marijuana Abuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Duke site has masked outcomes assessor; University of Connecticut site does not have masked outcomes assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MET/CBT-12 plus CBT-D (Experimental): CBT-D is an integrated cognitive behavior therapy targeting depression, delivered by the same study therapist who delivers MET/CBT-12 to the adolescent. All adolescents receiving CBT-D remain in MET/CBT-12 with their study provider.
  Interventions: Behavioral: MET/CBT-12; Behavioral: CBT-D
- MET/CBT-12 plus D-TAU (Active Comparator): D-TAU (Depression Treatment as Usual) consists of referral to a depression treatment provider in the community. In this study D-TAU will be enhanced by assistance from the study team in locating providers and, with consent, an assessment report about the adolescent from the study team to the provider. All adolescents receiving TAU for depression remain in MET/CBT-12 with their study provider.
  Interventions: Behavioral: MET/CBT-12; Other: D-TAU
- MET/CBT-12 alone (Active Comparator): MET/CBT-12 consists of two sessions of motivation enhancement therapy and 10 sessions of cognitive behavior therapy, targeting alcohol or cannabis abuse. All adolescents in the study receive MET/CBT-12 over 12 to 14 weeks.
  Interventions: Behavioral: MET/CBT-12

INTERVENTIONS:
Behavioral: MET/CBT-12 — Two sessions of motivation enhancement therapy followed by 10 sessions of cognitive behavior therapy targeting alcohol or cannabis abuse. These 12 sessions will be delivered over 12 to 14 weeks.
Behavioral: CBT-D — CBT-D consists of seven weekly sessions of cognitive behavior therapy targeting depression.
  Arms: MET/CBT-12 plus CBT-D
Other: D-TAU — D-TAU is treatment as usual in the community, targeting depression. It may consist of medication and/or behavioral intervention.
  Arms: MET/CBT-12 plus D-TAU

SUMMARY:
The investigators will recruit adolescents with alcohol or cannabis abuse and clinically significant depression. All participants will receive 12 sessions of an evidence-based treatment for alcohol abuse, Motivation Enhancement Therapy/Cognitive Behavior Therapy-12, over 12 to 14 weeks. Those who are still depressed after 4 weeks will be randomized to receive treatment augmentation with either an integrated cognitive behavior therapy for depression, delivered by their study therapist, or depression treatment-as-usual in the community. The study hypothesis is that integrated depression treatment will surpass community treatment-as-usual in efficacy.

DETAILED DESCRIPTION:
Alcohol and other substance use disorders (AOSUDs), primarily cannabis use disorders, continue to be a significant public health concern among American adolescents. AOSUDs are commonly accompanied by co-occurring psychiatric disorders including depression. This comorbidity has been associated with increased severity of AOSUD, earlier treatment termination, poorer outcomes, and increased suicidal risk. Presently there is neither a consensus nor a standard, evidence-based intervention to address the need for an effective and feasible treatment for both disorders. However, cognitive behavior therapy (CBT) has been found to be effective for each of these disorders, separately. In addition, in some, but not all, adolescents with both disorders, depression appears to respond rapidly to CBT that targets only alcohol or substance abuse. This suggests that early depression responders (EDRs) may not need additional treatment that targets depression directly, unlike their non-early responding (NEDR) counterparts. However, no studies have compared longer term outcomes of adolescent EDRs to NEDRs. Moreover, no randomized, controlled studies have tested the hypothesis that an integrated CBT intervention for co-occurring AOSUD and depression will be effective for both disorders, in NEDR adolescents.

In this two-site study, submitted in response to PA: PAS-10-251, we will recruit 170 eligible adolescents (102 at the University of Connecticut and 68 at Duke University), ages 13 years to 21 years-11 months, with alcohol or cannabis use disorders and clinically significant depression. All subjects will receive 12 sessions of Motivation Enhancement Therapy/Cognitive Behavior Therapy (MET/CBT-12), a standard, evidence-based intervention for alcohol or drug abuse over 12 to 14 weeks. After four weeks, NEDR adolescents will be randomized to depression treatment augmentation, either with seven sessions of CBT (CBT-D), integrated with MET/CBT-12, or with enhanced depression-treatment-as-usual in the community (D-ETAU). We estimate that 120 adolescents will be randomized; we will stratify randomization on gender, age, and presence/absence of a Major Depressive Episode. We will assess all 170 participants at baseline, weeks 4, 9, and 14 (after treatment), and at 3-, 6-, and 9-month follow-up.

The first aim of this study is to describe the percentage of depressed AOSUD adolescents who demonstrate EDR during alcohol or cannabis abuse treatment alone, examine EDR durability and EDR predictors. The second and third aims test the hypotheses that, for NEDR teens, an integrated treatment augmentation (CBT-D) will lead to better depression and alcohol or cannabis outcomes, respectively, than augmentation with D-ETAU. We will compare outcomes of all three groups (EDRs; and NEDRs in each augmentation), on alcohol use, depressive symptoms, alcohol- or cannabis-related functional impairment, maintenance of alcohol or cannabis treatment gains, and depression remission rates over time, and will analyze the temporal ordering of changes in alcohol or cannabis use and depression during and after treatment. This is the first study to test an adaptive treatment model with depressed alcohol or cannabis use disorder youths, and thus has significant potential to guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 years to 21 years, 11 months at baseline
* Current alcohol or cannabis abuse or dependence diagnosis (DSM-IV) OR current level of potentially harmful drinking or cannabis use as evidenced by (1) consumption of 4 or more drinks per drinking day (males) or three or more (females), or use of cannabis at least three times in past 90 days (or before admission into a controlled environment)
* Current clinically significant depression, defined as a score of 40 or more on the Children's Depression Rating Scale-Revised at baseline
* If currently taking anti-depressant medication, on a stable dose for at least one month
* Willingness to accept treatment
* Able to speak and read English (5th-grade level)
* Residence within 45-minute drive from treatment site
* Adolescent and a parent agree to sign Institutional Review Board approved consent/assent form; for subjects ages 18-19, parent involvement is optional and is the decision of the youth
* Parent/guardian agrees to provide collateral information and to designate two third parties who could be contacted in case the subject is lost to follow-up; for subjects ages 18-19, the participating youth will provide this information
* Participant (and parent, if youth is under age 18) not planning to move outside the area in the next 9 months.

Exclusion Criteria:

* Suicidal ideation with a plan, or suicide attempt within 30 days. In addition to such suicide risk being indicated in baseline interview material, a score exceeding the 89th percentile on the Suicide Ideation Questionnaire (SIQ-Jr), will necessitate an immediate risk assessment by the Independent Evaluator which may lead to exclusion under this criterion.
* Homicidal ideation with a plan or any plan to hurt others
* Lifetime diagnosis of psychosis, schizophrenia, bipolar disorder, intellectual disability or autistic disorder
* Current dependence on a substance other than alcohol, marijuana or nicotine
* Current non-alcohol or cannabis use disorder or depression primary diagnosis, i.e., the diagnosis requires care more urgently than does alcohol or cannabis use disorder or depression

Ages: 13 Years to 263 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2015-01-16 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Alcohol use frequency assessed with the Alcohol Consumption Questionnaire | Change from baseline to week 14; change from baseline to 9 months after treatment ends
  At every assessment point (baseline, weeks 4, 9, and 14 [end of treatment]; and then 3, 6, and 9 months after treatment ends, adolescents will be interviewed by an independent evaluator using the Alcohol Consumption Questionnaire regarding alcohol use frequency over the past three months (baseline, and months 3, 6, and 9) or past month (weeks 4, 9, and 14).
Severity of depression, as measured on the Children's Depression Rating Scale-Revised (CDRS-R) | Change from baseline to week 4; Change from baseline to week 14; Change from baseline to 9 months after treatment ends
  At every assessment point (baseline, weeks 4, 9, and 14 [end of treatment] and then 3, 6, and 9 months after treatment ends, adolescents and parents will be interviewed by an independent evaluator using the CDRS-R, with reference to the adolescent's depression symptoms during the past week. The week 4 assessment determines whether the adolescent is an early responder on depression, defined as having a 50% reduction in CDRS-R score. One item assesses suicidal thinking or behavior.
Alcohol use quantity assessed with the Alcohol Consumption Questionnaire | Change from baseline to week 14; Change from baseline to 9 months after treatment ends
  At every assessment point (baseline, weeks 4, 9, and 14 [end of treatment]; and then 3, 6, and 9 months after treatment ends, adolescents will be interviewed by an independent evaluator regarding alcohol use quantity over the past three months (baseline; months 3, 6, and 9) or past month (weeks 4, 9, and 14), using the Alcohol Consumption Questionnaire.
Cannabis use frequency assessed with the Drug Checklist | Change from baseline to week 14; Change from baseline to 9 months after treatment ends
  At every assessment point (baseline, weeks 4, 9, and 14 [end of treatment]; and then 3, 6, and 9 months after treatment ends, adolescents will be interviewed by an independent evaluator regarding cannabis use frequency over the past three months (baseline; months 3, 6, and 9) or past month (weeks 4, 9, and 14), using the Drug Checklist.

SECONDARY OUTCOMES:
Diagnosis | Baseline to Week 14; baseline to 9 Months after treatment ends
  At baseline, week 14 (end of treatment), and 9 months after treatment, the adolescent will complete the Voice DISC diagnostic interview to determine whether he or she continues to meet criteria for an alcohol or cannabis use disorder
Teen-Addiction Severity Index (T-ASI) | Baseline to Week 14; baseline to 9 months after treatment ends
  The Independent Evaluator will complete the T-ASI with the adolescent and parent at every assessment point (baseline, week 4, week 9, week 14, and then 3, 6, and 9 months after treatment ends) to determine whether there are changes in substance-use-related functional problems
Suicidal Ideation Questionnaire-Jr. High Version (SIQ-Jr) | Baseline to Week 14; baseline to 9 months after treatment ends
  Adolescents will complete this self-report form at every assessment point (baseline, week 4, week, 9, week 14; and then 3, 6, and 9 months after treatment ends) to determine if there are significant reductions in suicidal ideation
Children's Global Assessment of Functioning (CGAS) | Baseline to Week 14; baseline to 9 months after treatment ends
  The Independent Evaluator will make this single item rating of global functioning at every assessment point (baseline, week 4, week 9, week 14, and then 3, 6, and 9 months after treatment ends) to determine if there are significant improvements in adolescent's overall functioning
Clinical Global Impression-Improvement in Depression (CGI-I) | Baseline to Week 14; baseline to 9 months after treatment ends
  At every assessment point except baseline (at week 4, week 9, week 14, and then at 3, 6, and 9 months after treatment ends), the independent evaluator will rate the adolescent's improvement since baseline in the domain of depression, using CDRS-R scores as the reference. The CGI-I score determines whether the adolescent is a partial or full responder, or a non-responder to treatment.

OTHER OUTCOMES:
Beck Depression Inventory-II (BDI-II) | Baseline to Week 14; baseline to 9 months after treatment ends
  Adolescents will complete this self-report measure of depression severity at all assessment points (baseline, week 4, week 9, week 14; and then 3, 6, and 9 months after treatment ends) to determine if there has been a significant reduction in severity of depressive symptoms. One item assesses suicidal ideation or intent.
Situational Confidence Questionnaire (SCQ) | Baseline to Week 14
  At baseline, week 4, and week 14, the adolescent will self-report perceived self-efficacy to manage potentially stressful situations involving alcohol or cannabis, to determine if this confidence increases during treatment
Urine analysis | From baseline through month 9 of follow-up
  At every assessment point (baseline, week 4, week 9, week 14, and then 3, 6, and 9 months after treatment ends), and 8 additional times during treatment, adolescents will complete a 6-panel iCUP Drug Screen Test to check for non-alcohol substance use.

CONTACTS AND LOCATIONS:
Overall Officials: John F Curry, PhD, Principal Investigator — Duke University; Yifrah Kaminer, M.D., Principal Investigator — UConn Health
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Duke Child and Family Study Center, Durham, North Carolina

REFERENCES:
- [Derived] Curry JF, Kaminer Y, Goldston DB, Chan G, Wells KC, Burke RH, Inscoe AB, Meyer AE, Cheek SM. Adaptive Treatment for Youth With Substance Use and Depression: Early Depression Response and Short-term Outcomes. J Am Acad Child Adolesc Psychiatry. 2022 Apr;61(4):508-519. doi: 10.1016/j.jaac.2021.07.807. Epub 2021 Aug 6. PMID 34371102